CLINICAL TRIAL: NCT02341443
Title: A Multicenter Randomized Controlled Clinical Investigation to Investigate the Treatment of Double (Bilateral) Mandibular Fractures
Brief Title: A Multicenter RCT to Investigate the Treatment of Double (Bilateral) Mandibular Fractures
Acronym: DMFx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: AOCMF (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP_DMFx_V1.0
Record Dates: First submitted 2014-12-04; First posted 2015-01-19 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Mandibular Fractures
Keywords: bilateral double mandibular fractures; rigid fixation; no-rigid fixation; jaw
MeSH Terms: conditions — Mandibular Fractures | interventions — Drug Implants; Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rigid (Experimental): Surgery using mandibulo-maxillary fixation, implants providing rigid fixation on most anterior fracture and non-rigid fixation on the most posterior fracture.
  Interventions: Procedure: Implants
- Non-rigid (Active Comparator): Surgery using mandibulo-maxillary fixation and implants providing non-rigid fixation on both fracture sides.
  Interventions: Procedure: Implants

INTERVENTIONS:
Procedure: Implants — Experimental arm: Rigid
  Surgical treatment using arch bars and according to the following fixation:
  Rigid fixation on one side (most anterior fracture) and non-rigid fixation on the other (most posterior fracture).
  Active comparator: Non-rigid
  Surgical treatment using arch bars and according to the following fixation:
  Non-rigid fixation on both fracture sides.
  Whereas non-rigid fixation is defined as a single miniplate of ≤1.00 mm thickness, and rigid fixation is defined as a single plate of ≥1.25 mm thickness, a combination of 2 plates or a 3D geometric plate.
  Other Names: Open reduction and internal fixation

SUMMARY:
Mandibular fractures represent approximately 50% of the total facial fractures and are commonly (more than half) presented in more than one location. A few simple fractures can be treated using a conservative approach. More often, however, mandibular fractures require stabilization using open reduction and internal fixation.

Simple mandibular fractures can be treated using non-rigid fixation techniques that rely on the load-sharing principle, by which stabilization is accomplished with both fixation devices and bone surfaces. On the other hand, more complex fractures with continuity defects or comminuted need to be handle using rigid fixation where the device assumes all the forces (load-bearing principle). These approaches are well established, whereas the level of evidence for the treatment of bilateral double mandibular fractures (DMF) is still scarce. In fact, which surgical treatment, or combination of treatments, leads to the best outcome and the lowest rate of complications in bilateral DMFs is an open question.

The purpose of this study is to assess the complication rate in patients suffering from bilateral DMF treated either using non-rigid fixation on both fracture sides or a combination of rigid fixation on one side and non-rigid fixation on the other side.

DETAILED DESCRIPTION:
Prospective data will be collected in 314 patients suffering from bilateral (double) mandibular fracture randomly treated either with non-rigid fixation on both fracture sides or a combination of rigid fixation on one side and non-rigid fixation on the other side. This is a study where patients will be treated per randomization to one of the two established treatments and followed for further clinical examination post-operatively at 6 weeks and 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the date of the surgery
* Diagnosis of bilateral (double) mandibular fracture located in:

  * Angle and body or
  * Angle and symphysis or
  * Body and symphysis
* Dentition: Patients must have most of their maxillary and mandibular teeth present and it must be possible to identify proper occlusion. The application of intraoperative Mandibulo-maxillary fixation (MMF) using arch bars must be possible
* Ability to understand the content of the patient information / Informed Consent Form
* Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
* Signed and dated IRB/EC-approved written informed consent

Exclusion Criteria:

* Fractures displaying continuity defect or comminution
* Fractures showing clinical signs of infection at presentation
* Edentulous mandible fracture
* Fractures requiring an extra-oral surgical approach
* Concomitant maxillary fractures
* Concomitant condylar fracture
* Prior surgical treatment of the mandibular fracture(s)
* Atrophy of the mandible (<20 mm vertical height) at the level of the fracture(s)
* Polytrauma (i.e. severe injuries leading to life-threatening condition)
* Prisoners
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2015-04; Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of anticipated procedure- or condition-related Adverse Events | 6 weeks

SECONDARY OUTCOMES:
Degree of displacement of the fracture | Pre-operatively (Day -1)
Location of the tooth with respect to the line of fracture | Pre-operatively (Day -1)
Mechanism of production of the fracture: | Pre-operatively (Day -1)
Time in days between the occurrence of the injury and the surgery | Intraoperatively (Day 0)
Length of the surgery | Intraoperatively (Day 0)
  Time in minutes from the first incision to skin closure
Length of the hospital stay | Intraoperatively (Day 0)
  Time in days between the admission and the discharge of the (acute) hospital
Characteristics of the hardware | Intraoperatively (Day 0)
  Characteristics of the hardware/device used to reduce the fracture concerning its shape, thickness and number or screws
Use of antibiotics | Intraoperatively (Day 0)
  Administration of antibiotics during surgery
Difficulty of application of the hardware | Intraoperatively (Day 0)
  Surgeon's own assessment of difficulty of application of the hardware from very easy to very difficult
Dysfunction of the mandible | 6 weeks, 3 months
  Helkimo Index

CONTACTS AND LOCATIONS:
Overall Officials: Risto Kontio, MD DDS PhD, Principal Investigator — Helsinki University Central Hospital; Edward Ellis III, DDS MS, Principal Investigator — UT Health Science Center at San Antonio
Locations (11):
- United States (2):
  - Jacobi Medical Center, New York, New York
  - UT Health Science Center at San Antonio, San Antonio, Texas
- Helsinki University Hospital, Helsinki, Finland
- Germany (2):
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Ludwig-Maximillians University, München
- Hospital Sg Buloh, Sungai Buloh, Malaysia
- Hamad Medical Corporation, Doha, Qatar
- Emergency Clinical County Hospital of Constanta, Constanța, Romania
- King Edward VIII Hospital, Durban, South Africa
- 12 de Octubre University Hospital, Madrid, Spain
- Lviv Regional Clinical Hospital (Lviv National Medical University), Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rughubar V, Vares Y, Singh P, Filipsky A, Creanga A, Iqbal S, Alkhalil M, Kormi E, Hanken H, Calle AR, Smolka W, Turner M, Csaki G, Sanchez-Aniceto G, Perez D, Cornelius CP, Alani B, Vlad D, Kontio R, Ellis E 3rd. Combination of Rigid and Nonrigid Fixation Versus Nonrigid Fixation for Bilateral Mandibular Fractures: A Multicenter Randomized Controlled Trial. J Oral Maxillofac Surg. 2020 Oct;78(10):1781-1794. doi: 10.1016/j.joms.2020.05.012. Epub 2020 May 15. PMID 32589939